CLINICAL TRIAL: NCT03296735
Title: A Difference in the Cross-section Area of Subclavian Vein Between Supine and Lateral Tilt Position: Its Clinical Impact on Subclavian Venous Catheterization - Stage II
Brief Title: A Difference in Subclavian Vein Catheterization Between Supine and Lateral Tilt Position - Stage I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-110-871-1
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Catheterization; Posture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ipsilateral tilt (Experimental): Measuring the cross-sectional area of right subclavian vein in the 20 degree left tilting posture.
  Interventions: Procedure: Ipsilateral tilt
- Supine (No Intervention): Measuring the cross-sectional area of right subclavian vein in supine position.
- Contralateral tilt (Active Comparator): Measuring the cross-sectional area of right subclavian vein in the 20 degree left tilting posture.
  Interventions: Procedure: Contralateral tilt

INTERVENTIONS:
Procedure: Ipsilateral tilt — The operation table will be tilted 20 degrees right laterally.
  Arms: Ipsilateral tilt
Procedure: Contralateral tilt — The operation table will be tilted 20 degrees left laterally.
  Arms: Contralateral tilt

SUMMARY:
Central venous catheterization is widely used for various purposes during surgery. For central venous catheterization, subclavian vein is selected because of the relatively low risk of infection, long-term patency and low patient discomfort. The cross - sectional area of the subclavian vein is an important factor to increase success rate. Several studies have reported that the Trendelenburg position increases the cross-sectional area of the subclavian vein, and the lateral tilt position can change the cross-sectional area of the subclavian vein. However, the impact of lateral tilt position to the cross-sectional area of the subclavian vein is not clear. The ipsilateral position can increase the cross-sectional area of the subclavian vein, and the contralateral position can decrease the cross-sectional area by gravity.

In the first stage of this study, we compare the cross-sectional area of subclavian vein using ultrasonography in supine, ipsilateral, and contralateral tilt position.

ELIGIBILITY:
Inclusion Criteria:

- the patients who receive elective neurosurgical surgery and require central venous catheter

Exclusion Criteria:

* the patients who have puncture site infection
* the patients who have chemoport, pacemaker in right subclavian vein
* the patients who had received right mastectomy or right pneumonectomy
* other contraindications for subclavian venous catheterization (eg. mass, hematoma, vegetation, and anticoagulation)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2017-10-15 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The cross-sectional area of right subclavian vein | 1 minutes after position change
  The cross-sectional area of right subclavian vein

REFERENCES:
- [Derived] Yoon HK, Lee HC, Kang P, Lee JM, Park HP, Cho YJ. Effects of ipsilateral tilt position on the cross-sectional area of the subclavian vein and the clinical performance of subclavian vein catheterization: a prospective randomized trial. BMC Anesthesiol. 2020 Sep 5;20(1):226. doi: 10.1186/s12871-020-01144-1. PMID 32891115
- [Derived] Jung DE, Lee HC, Yoon HK, Park HP. The effects of ipsilateral tilt position on right subclavian venous catheterization: study protocol for a prospective randomized trial. Trials. 2018 May 24;19(1):292. doi: 10.1186/s13063-018-2666-8. PMID 29793550